CLINICAL TRIAL: NCT07121855
Title: Symptoms and Coping Strategies Among Patients With Implantable Cardioverter Defibrillators
Brief Title: Symptoms and Coping Strategies Among Patients With Implantable Cardioverter Defibrillator
Acronym: ICD
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sebiha Aktaş Us, Nurse Specialist, TC Erciyes University
Other Study IDs: Adana
Record Dates: First submitted 2025-08-02; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Sudden Cardiac Arrest; Ventricular Arrhythmias
Keywords: Implantable Defibrillators; Symptoms; Self Care; Arrhythmias; Symptom Management
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with implantable cardioverter defibrillators (ICDs): Patients who have had an implantable cardioverter defibrillator (ICD) implanted at least 3 months prior

SUMMARY:
Implantable cardioverter defibrillators (ICDs) are widely used to prevent sudden cardiac death in patients with serious arrhythmias and significantly increase survival rates. However, living with an ICD can bring about a range of physical symptoms, such as palpitations, fatigue, and chest discomfort, as well as psychological challenges like anxiety, fear of shock, and uncertainty about the future. These symptoms can negatively impact patients' quality of life and daily functioning. As a result, how patients cope with these experiences becomes an important component of long-term well-being. Despite advancements in device technology, many patients continue to experience emotional and behavioral adjustment challenges. Researching patients' symptom experiences and coping strategies is essential for developing supportive, non-pharmacological interventions that address both physical and emotional needs. This study aims to identify the most common symptoms associated with ICD and investigate the methods patients use to manage them in their daily lives.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillators (ICDs) are widely used medical devices designed to prevent sudden cardiac death in patients with life-threatening ventricular arrhythmias. Although ICD therapy has significantly improved survival rates in high-risk heart patients, its presence can introduce new physical and psychological challenges that may impact daily life. Patients living with an ICD often report various symptoms such as palpitations, fatigue, chest discomfort, and sleep disturbances. In addition to these physical symptoms, psychological distress such as anxiety, fear of shock, and uncertainty about the future is also commonly observed.

Transitioning to life with an ICD requires not only physiological adaptation but also emotional and behavioral adjustment. How patients perceive the presence of the device and how they cope with it plays a critical role in their overall quality of life. While technological advancements have reduced inappropriate shocks and device-related complications, the psychosocial burden remains significant for many patients. As a result, coping strategies, particularly non-pharmacological approaches, have become essential tools for managing stress associated with ICDs and maintaining psychological balance.

Despite the increasing number of ICD recipients, there remains a gap in the literature regarding the specific symptoms experienced post-implantation and the individual coping mechanisms employed by patients. Investigating these dimensions could provide healthcare providers with insights into the ongoing needs of ICD patients and guide the development of supportive interventions that address both physical symptoms and emotional responses.

This study aims to identify the most common symptoms among ICD patients and investigate the methods they use to cope with these symptoms. By better understanding patient experiences, clinicians can provide more comprehensive and patient-centered care tailored to this unique population.

ELIGIBILITY:
Inclusion Criteria:

* Participants were informed about the study and provided informed consent to participate voluntarily,
* Patients who had an ICD implanted at least 3 months prior to the study,
* Patients with no communication difficulties (speak Turkish, no mental retardation),
* Adult patients aged 18 years or older.

Exclusion Criteria:

* Patients who are unable to provide informed consent regarding the study
* Patients who have undergone ICD implantation less than 3 months prior
* Patients who have difficulty communicating
* Patients under the age of 18
* Patients whose symptoms cannot be directly attributed to the ICD due to serious physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD patients
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Types and frequencies of symptoms | Baseline
  Types and frequencies of physical and psychological symptoms reported by patients with implantable cardioverter defibrillator (ICDs)
Types and frequencies of coping strategies | Baseline
  Types and frequencies of coping strategies used by ICD patients to manage their symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Taşcı, Professor, Study Director — TC Erciyes University
Locations (1):
- Turkish Ministry of Health, Adana City Training and Research Hospital, Sinop, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Not applicable. No individual participant data (IPD) will be shared.

REFERENCES:
- [Background] Polikandrioti M, Tzirogiannis K, Zyga S, Gerogianni G, Stefanidou S, Tsami A, Panoutsopoulos G. Assessment of fatigue in patients with a permanent cardiac pacemaker: prevalence and associated factors. Arch Med Sci Atheroscler Dis. 2018 Dec 20;3:e166-e173. doi: 10.5114/amsad.2018.81085. eCollection 2018. PMID 30775608
- [Background] Polikandrioti M, Tzirogiannis K, Zyga S, Koutelekos I, Vasilopoulos G, Theofilou P, Panoutsopoulos G. Effect of anxiety and depression on the fatigue of patients with a permanent pacemaker. Arch Med Sci Atheroscler Dis. 2018 Feb 5;3:e8-e17. doi: 10.5114/amsad.2018.73231. eCollection 2018. PMID 30775584
- [Background] Pasyar N, Rambod M, Nikoo MH, Mansouri P. An Evaluation of the Association between Quality of Life and Psychological Issues in Patients with Automated Implantable Cardioverter Defibrillator. J Caring Sci. 2021 Nov 6;11(1):28-35. doi: 10.34172/jcs.2022.01. eCollection 2022 Mar. PMID 35603084
- [Background] Magnusson P, Mattsson G, Wallhagen M, Karlsson J. Health-related quality of life in patients with implantable cardioverter defibrillators in Sweden: a cross-sectional observational trial. BMJ Open. 2021 Jul 9;11(7):e047053. doi: 10.1136/bmjopen-2020-047053. PMID 34244266
- [Background] Sun Y, Yu Z. Anxiety and depression in a patient with an implantable cardioverter defibrillator for early repolarization syndrome: A case report and clinical discussion. Journal of Clinical and Basic Psychosomatics. 2024;2(3):2848.
- [Background] Rambod M, Rohaninasab S, Pasyar N, Nikoo MH. The effect of virtual interactive nurse-led support group intervention on fatigue, shock anxiety, and acceptance of implantable cardioverter defibrillator patients: a randomized trial. BMC Cardiovasc Disord. 2024 Jan 11;24(1):40. doi: 10.1186/s12872-024-03713-5. PMID 38212701
- [Background] Spar DS, Bianco NR, Knilans TK, Czosek RJ, Anderson JB. The US Experience of the Wearable Cardioverter-Defibrillator in Pediatric Patients. Circ Arrhythm Electrophysiol. 2018 Jul;11(7):e006163. doi: 10.1161/CIRCEP.117.006163. PMID 29945928
- [Background] Sert, M. (2019). İpmplante edilebilir kardiyoverter defibrilatörü olan hastalarda ölüm kaygısı ve uyku kalitesi. Turk J Cardiovasc Nurs 2019;10(22):78-86.
- [Background] da Silva KR, Costa R, Rodrigues CG, Schasechter A, Nobre MC, Passman R, Mark DB. Quality of life in patients with implantable cardioverter-defibrillator: systematic review of randomized controlled trials. Eur J Cardiovasc Nurs. 2018 Mar;17(3):196-206. doi: 10.1177/1474515117739619. Epub 2017 Oct 25. PMID 29067836
- [Background] Bozat A.D. (2019). Kalp İçi Defibrillatör Ve Kalıcı Kalp Pili Kullanan Çocuk, Ergen Ve Ailelerinde Dayanıklılık, Yaşam Kalitesi Ve Psikiyatrik Semptomların Değerlendirilmesi. (Uzmanlık Tezi, Hacettepe Üniversitesi Tıp Fakültesi Çocuk Sağlığı Ve Hastalıkları Anabilim Dalı).
- [Background] Forman J, Baumbusch J, Jackson H, Lindenberg J, Shook A, Bashir J. Exploring the patients' experiences of living with a subcutaneous implantable cardioverter defibrillator. Eur J Cardiovasc Nurs. 2018 Dec;17(8):698-706. doi: 10.1177/1474515118777419. Epub 2018 May 18. PMID 29775072